CLINICAL TRIAL: NCT05140343
Title: Effectiveness of Mobile Electrocardiogram Monitoring for Detecting Arrhythmias in Children With Symptoms: A Randomized Clinical Trial
Brief Title: Mobile Electrocardiogram Monitoring for Detecting Arrhythmias in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Section, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SMART-CHILD
Record Dates: First submitted 2021-08-08; First posted 2021-12-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Arrhythmias, Cardiac; Children, Only; Congenital Heart Disease; Sudden Cardiac Death; Diagnoses Disease
Keywords: grown ups with congenital heart (GUCH) disease; pediatric cardiology; diagnosis of arrhythmia; new diagnostic tools; early diagnosis; prevention
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Defects, Congenital; Death, Sudden, Cardiac; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile ECG Monitoring (Experimental): Standard care with clinical follow-up plus Mobile ECG Monitoring.
  Interventions: Diagnostic Test: KARDIA Mobile ECG Monitoring (KMCM)
- 24-hour Holter monitoring (No Intervention): Standard care with clinical follow-up plus repeating 24-hours Holter ECG (month 1, 6, 12)

INTERVENTIONS:
Diagnostic Test: KARDIA Mobile ECG Monitoring (KMCM) — The KMCM will be introduced to the patient of the KMCM arm in the outpatient clinic. The activation and configuration will be done together with the physician in the outpatient clinic (installation of the ECG app, enabling heart rate rhythm notification). Patients are requested to acquired ECGs twice weekly plus additional ECGs if symptomatic. In case of symptoms the patient is asked to generate an ECG and communicate the event timely to the investigator and to the treating physician by sending a report through the ECG app. An e-mail account created for the study will be checked at least once a day. The arrhythmia diagnosis will be performed by the clinician based on the ECG information, independently of the arrhythmia classification automatically performed by the device. In case of stronger symptoms of any kind at any time the patient is asked to request medical help regardless of the KMCM notifications. Change of management will be collected.
  Arms: Mobile ECG Monitoring

SUMMARY:
The objective of this project is to evaluate the capability of a specific mobile electrocardiogram monitoring of detecting arrhythmic events in children with history of palpitation and or syncope. We will compare this approach with the standard approach of clinical follow-up plus 24-hour Holter ECG monitoring in terms of acceptability and ability to identify significant arrhythmias.

DETAILED DESCRIPTION:
Syncope and palpitation are one of the most common referrals to pediatric cardiology in patients with and without structural heart disease. In children with palpitation supraventricular tachycardia (SVT) is the most common final diagnosis. While some SVTs caused by the presence of an accessory pathway are highly recommend to be treated, other forms of arrhythmia are rarely life threatening and therapy depends on the burden of symptoms. Some SVT can be the first manifestation of an underlying heart disease. Early onset of atrial fibrillation, for example, in childhood usually reveals a genetic pathology and therefore needs further investigation. Besides the need for precise diagnosis to choose adequate management and therapy, unrecognized paroxysmal SVT have shown to lead to misdiagnosis mimicking symptoms of a psychiatric disorder. However, with the current diagnostic tools and protocols in only 10 % to 15 % of children with palpitation an underlying arrhythmia is found.

Syncope commonly is of benign character in children but it can be the first warning sign of a serious condition. Despite considerable testing and expense accurate diagnosis of the underlying cause of syncope is still challenging. The theoretical possibility of an underlying fatal arrhythmia adds remarkable to the mental health challenges of adolescence and the families. Sudden cardiac death (SCD) is a rare but devastating event in children and adolescents.

Syncope and palpitation deserve even higher attention in patients with congenital heart disease (CHD). These patients have an overall higher risk of developing cardiac arrhythmias as consequence of the pre-existing anatomical alterations, as well as the surgical treatment necessary for its correction. In many cases arrhythmia occur earlier in life and sometimes SCD is the first symptom of manifestation.

To study the origin of palpitation and syncope 12 lead electrocardiogram (ECG) and 24-hours Holter monitoring is typically performed. In case of high clinical suspicion, implantable loop-recorder and electrophysiological study can be performed to finally reach a diagnosis. However, it is an invasive test that is thought to be avoided in children if possible and might be poorly tolerated in patients with CHD.

In recent years, technological development has allowed the validation of different tools for detection of arrhythmias by "smart" devices. The "KARDIA" Mobile Cardiac Monitor is a handheld ECG device that enables users to collect and store single-channel ECG recordings using the smart phone, smart watch, or tablet. A recent study has demonstrated the efficacy of this device in the early diagnosis of arrhythmic disorders in adults by performing ECGs twice weekly plus additional ECG if symptomatic. However, its utility for the early detection and diagnosis of arrhythmias in children and patients with a CHD, which have a different normal physiology of the heart rhythm, has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-18 years old with or without the diagnosis of structural heart disease and symptoms suggestive of rhythm disorders as follows: palpitations and/or syncope and/or dizziness.
* 24-hours Holter without diagnosis of arrhythmia.
* Having an smart phone, smart watch, or tablet (the patient itself or a family member who lives together with the patient) compatible with KARDIA mobile ECG monitoring.
* Signed informed consent. In cases under the age of <18 y.o informed consent should be signed by parents or guardians.

Exclusion Criteria:

* Concomitant investigation treatments.
* Being already diagnosed for arrhythmic events.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent.
* Patient's refusal to participate in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to a documented new arrhythmia. | 12 months
  Time to a documented new arrhythmia counting time from the inclusion date.

SECONDARY OUTCOMES:
Incidence of medical request | 12 months
  Rate of patients with changes of diagnostic and/or therapy
Hospitalization during study time. | 12 months
  Number of participants hospitalized during study time

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Médico Teknon
Locations (1):
- Centro Medico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherwin ED, Berul CI. Sudden Cardiac Death in Children and Adolescents. Card Electrophysiol Clin. 2017 Dec;9(4):569-579. doi: 10.1016/j.ccep.2017.07.008. PMID 29173403
- [Background] Buddhe S, Singh H, Du W, Karpawich PP. Radiofrequency and cryoablation therapies for supraventricular arrhythmias in the young: five-year review of efficacies. Pacing Clin Electrophysiol. 2012 Jun;35(6):711-7. doi: 10.1111/j.1540-8159.2012.03372.x. Epub 2012 Mar 27. PMID 22452328
- [Background] Pappone C, Manguso F, Santinelli R, Vicedomini G, Sala S, Paglino G, Mazzone P, Lang CC, Gulletta S, Augello G, Santinelli O, Santinelli V. Radiofrequency ablation in children with asymptomatic Wolff-Parkinson-White syndrome. N Engl J Med. 2004 Sep 16;351(12):1197-205. doi: 10.1056/NEJMoa040625. PMID 15371577
- [Background] McCrank E, Schurmans K, Lefcoe D. Paroxysmal supraventricular tachycardia misdiagnosed as panic disorder. Arch Intern Med. 1998 Feb 9;158(3):297. doi: 10.1001/archinte.158.3.297. No abstract available. PMID 9472212
- [Background] Sedaghat-Yazdi F, Koenig PR. The teenager with palpitations. Pediatr Clin North Am. 2014 Feb;61(1):63-79. doi: 10.1016/j.pcl.2013.09.010. Epub 2013 Oct 12. PMID 24267458
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] MacCormick JM, McAlister H, Crawford J, French JK, Crozier I, Shelling AN, Eddy CA, Rees MI, Skinner JR. Misdiagnosis of long QT syndrome as epilepsy at first presentation. Ann Emerg Med. 2009 Jul;54(1):26-32. doi: 10.1016/j.annemergmed.2009.01.031. Epub 2009 Mar 12. PMID 19282063
- [Background] Johnson ER, Etheridge SP, Minich LL, Bardsley T, Heywood M, Menon SC. Practice variation and resource use in the evaluation of pediatric vasovagal syncope: are pediatric cardiologists over-testing? Pediatr Cardiol. 2014 Jun;35(5):753-8. doi: 10.1007/s00246-013-0848-4. Epub 2013 Dec 17. PMID 24343729
- [Background] Sheldon R. Syncope outcomes in a national health database: low risk is not no risk. J Am Coll Cardiol. 2013 Jan 22;61(3):333-4. doi: 10.1016/j.jacc.2012.10.019. Epub 2012 Dec 12. No abstract available. PMID 23246387
- [Background] Nakano Y, Wataru S. Syncope in patients with inherited arrhythmias. J Arrhythm. 2017 Dec;33(6):572-578. doi: 10.1016/j.joa.2017.07.007. Epub 2017 Oct 6. PMID 29255503
- [Background] Longmuir PE, Sampson M, Ham J, Weekes M, Patel BJ, Gow RM. The mental health of adolescents and pre-adolescents living with inherited arrhythmia syndromes: a systematic review of the literature. Cardiol Young. 2018 May;28(5):621-631. doi: 10.1017/S104795111700289X. Epub 2018 Jan 18. PMID 29345602
- [Background] von Alvensleben JC. Syncope and Palpitations: A Review. Pediatr Clin North Am. 2020 Oct;67(5):801-810. doi: 10.1016/j.pcl.2020.05.004. Epub 2020 Aug 11. PMID 32888682
- [Background] Sliwa K, Azibani F, Johnson MR, Viljoen C, Baard J, Osman A, Briton O, Ntsekhe M, Chin A. Effectiveness of Implanted Cardiac Rhythm Recorders With Electrocardiographic Monitoring for Detecting Arrhythmias in Pregnant Women With Symptomatic Arrhythmia and/or Structural Heart Disease: A Randomized Clinical Trial. JAMA Cardiol. 2020 Apr 1;5(4):458-463. doi: 10.1001/jamacardio.2019.5963. PMID 32074256
- [Background] Brouwer C, Hazekamp MG, Zeppenfeld K. Anatomical Substrates and Ablation of Reentrant Atrial and Ventricular Tachycardias in Repaired Congenital Heart Disease. Arrhythm Electrophysiol Rev. 2016 Aug;5(2):150-60. doi: 10.15420/AER.2016.19.2. PMID 27617095
- [Background] Koyak Z, de Groot JR, Bouma BJ, Zwinderman AH, Silversides CK, Oechslin EN, Budts W, Van Gelder IC, Mulder BJ, Harris L. Sudden cardiac death in adult congenital heart disease: can the unpredictable be foreseen? Europace. 2017 Mar 1;19(3):401-406. doi: 10.1093/europace/euw060. PMID 27247006
- [Background] Motonaga KS, Khairy P, Dubin AM. Electrophysiologic therapeutics in heart failure in adult congenital heart disease. Heart Fail Clin. 2014 Jan;10(1):69-89. doi: 10.1016/j.hfc.2013.09.011. PMID 24275296
- [Background] Gourraud JB, Khairy P, Abadir S, Tadros R, Cadrin-Tourigny J, Macle L, Dyrda K, Mondesert B, Dubuc M, Guerra PG, Thibault B, Roy D, Talajic M, Rivard L. Atrial fibrillation in young patients. Expert Rev Cardiovasc Ther. 2018 Jul;16(7):489-500. doi: 10.1080/14779072.2018.1490644. Epub 2018 Jul 2. PMID 29912584
- [Background] Crawford MH, Bernstein SJ, Deedwania PC, DiMarco JP, Ferrick KJ, Garson A Jr, Green LA, Greene HL, Silka MJ, Stone PH, Tracy CM, Gibbons RJ, Alpert JS, Eagle KA, Gardner TJ, Gregoratos G, Russell RO, Ryan TH, Smith SC Jr. ACC/AHA Guidelines for Ambulatory Electrocardiography. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the Guidelines for Ambulatory Electrocardiography). Developed in collaboration with the North American Society for Pacing and Electrophysiology. J Am Coll Cardiol. 1999 Sep;34(3):912-48. doi: 10.1016/s0735-1097(99)00354-x. No abstract available. PMID 10483977
- [Background] Halcox JPJ, Wareham K, Cardew A, Gilmore M, Barry JP, Phillips C, Gravenor MB. Assessment of Remote Heart Rhythm Sampling Using the AliveCor Heart Monitor to Screen for Atrial Fibrillation: The REHEARSE-AF Study. Circulation. 2017 Nov 7;136(19):1784-1794. doi: 10.1161/CIRCULATIONAHA.117.030583. Epub 2017 Aug 28. PMID 28851729